CLINICAL TRIAL: NCT05974267
Title: Phase 2a Proof-of-Concept, Multicenter, Randomized, Open Label Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of a Single Dose of the Combination M5717-pyronaridine as Chemoprevention in Asymptomatic Adults and Adolescents With Plasmodium Falciparum Malaria Infection (CAPTURE-2)
Brief Title: Efficacy, Safety, and PK of M5717 in Combination With Pyronaridine as Chemoprevention in Adults and Adolescents With Asymptomatic Plasmodium Falciparum Infection (CAPTURE-2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201618_0034
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Malaria Infection
Keywords: Plasmodium falciparum; Chemoprevention; Malaria; Plasmodium eukaryotic translation elongation factor 2 (PeEF2); Exposure response; Adults; Adolescents; Asymptomatic Infection
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Asymptomatic Infections | interventions — pyronaridine; atovaquone, proguanil drug combination

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: M5717 (60 mg) + Pyronaridine (Experimental): Participants received single oral dose of M5717 60 milligram (mg) plus pyronaridine tetraphosphate (pyronaridine) 720 mg (Participants >= 65 kilogram [kg]) or pyronaridine 540 mg (Participants >= 45 to < 65 kg) once daily in a single day treatment regimen.
  Interventions: Drug: M5717 60 mg; Drug: Pyronaridine
- Cohort 2: M5717 (200 mg) + Pyronaridine (Experimental): Participants received single oral dose of M5717 200 mg plus pyronaridine 720 mg (Participants >= 65 kg) or pyronaridine 540 mg (Participants >= 45 to < 65 kg) once daily in a single day treatment regimen.
  Interventions: Drug: Pyronaridine; Drug: M5717 200 mg
- Cohort 3: M5717 (660 mg)+ Pyronaridine (Experimental): Participants received single oral dose of M5717 660 mg plus pyronaridine 720 mg (Participants >= 65 kg) or pyronaridine 540 mg (Participants >= 45 to < 65 kg) once daily in a single day treatment regimen.
  Interventions: Drug: Pyronaridine; Drug: M5717 660mg
- Cohort 4: Atovaquone-proguanil (Experimental): Participants received orally 3 doses of Malarone (fixed-dose combination of atovaquone-proguanil) once daily in a 3-day treatment regimen.
  Interventions: Drug: Atovaquone-Proguanil

INTERVENTIONS:
Drug: M5717 60 mg — Participants received single oral dose (Capsules) of 60 mg M5717 on Day 1 under fasting condition
  Arms: Cohort 1: M5717 (60 mg) + Pyronaridine
Drug: Pyronaridine — Participants received Pyronaridine tablets orally single dose of 720 (Participants >= 65 kg) and 540 mg (Participants >= 45 to < 65 kg) on Study Day 1 under fasting condition
  Other Names: Pyronaridine tetraphosphate
  Arms: Cohort 1: M5717 (60 mg) + Pyronaridine; Cohort 2: M5717 (200 mg) + Pyronaridine; Cohort 3: M5717 (660 mg)+ Pyronaridine
Drug: Atovaquone-Proguanil — Participants received Atovaquone-Proguanil tablets 1000/400 mg once daily in a 3-day treatment regimen.
  Arms: Cohort 4: Atovaquone-proguanil
Drug: M5717 200 mg — Participants received single oral dose (Capsules) of 200 mg M5717 on Day 1 under fasting condition
  Arms: Cohort 2: M5717 (200 mg) + Pyronaridine
Drug: M5717 660mg — Participants received single oral dose (Capsules) of 660 mg M5717 on Day 1 under fasting condition
  Arms: Cohort 3: M5717 (660 mg)+ Pyronaridine

SUMMARY:
This study evaluates the efficacy and safety of a single dose of M5717 plus pyronaridine tetraphosphate in clearing current Plasmodium falciparum infection and protecting against recurrent infections in asymptomatic adults and adolescents. The study will also assess the duration of protection provided by different doses of M5717 plus pyronaridine and the additional contribution of M5717 to the duration of protection using external study data.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Asymptomatic Plasmodium falciparum Malaria with no Fever or other sign of Acute Uncomplicated Malaria and, with Microscopic confirmation using Giemsa-stained thick film, and a Parasitemia of >= 40 to <= 10,000 Asexual Parasites/Microliter (μL) of Blood.
* Axillary Temperature < 37.0 degree Celcius (ºC) or oral/Tympanic/rectal Temperature< 37.5ºC; without history of fever during the previous 48 hours.
* Have a body weight >= 45 kilogram (kg)
* Participants capable of giving Signed Informed consent which includes Compliance with the requirements and restriction listed in the Informed consent form
* Other Protocol defined Inclusion Criteria could apply

Exclusion Criteria:

* Participants with any disease requiring Chronic Treatment
* Participants with any Preplanned surgery during the study
* Participants with any previous Treatment with pyronaridine as part of a combination therapy during the last 3 months
* Participants with any adequate Hematological, Hepatic, and renal function as defined in the Protocol
* Other protocol defined Exclusion Criteria could apply

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 192 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2024-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (4):
- Groupe de Recherche Action en Sante (GRAS), Ouagadougou, Burkina Faso
- Kisumu County Referral Hospital, Kisumu, Kenya
- MRC Unit The Gambia at LSHTM, Banjul, The Gambia
- Ndola Teaching Hospital, Ndola, Zambia

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=ms201618_0034
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: M5717 (60 mg) + Pyronaridine: Participants received a single oral dose of M5717 60 milligrams (mg) plus pyronaridine tetraphosphate (pyronaridine) 720 mg (for participants more than equal to (≥) 65 kilograms [kg]) or pyronaridine 540 mg (for participants ≥ 45 to less than (<) 65 kg) once daily in a single-day treatment regimen on Day 1 under fasting condition.
- Cohort 2: M5717 (200 mg) + Pyronaridine: Participants received a single oral dose of M5717 200 milligrams (mg) along with pyronaridine tetraphosphate (pyronaridine)-either 720 mg for those weighing ≥ 65 kilograms (kg) or 540 mg for those weighing between ≥ 45 kg and < 65 kg-in a single-day treatment regimen administered under fasting conditions on Day 1 under fasting condition.
- Cohort 3: M5717 (660 mg)+ Pyronaridine: participants received a single oral dose of M5717 660 mg along with pyronaridine-either 720 mg for those weighing ≥ 65 kilograms (kg) or 540 mg for those weighing between ≥ 45 kg and < 65 kg-as part of a single-day treatment regimen on Day 1 under fasting condition.
- Cohort 4: Atovaquone-proguanil: Participants received three oral doses of Malarone-a fixed-dose combination of 1000 mg atovaquone and 400 mg proguanil-administered once daily over a 3-day treatment regimen.
Period: Overall Study
Arm/Group | Cohort 1: M5717 (60 mg) + Pyronaridine | Cohort 2: M5717 (200 mg) + Pyronaridine | Cohort 3: M5717 (660 mg)+ Pyronaridine | Cohort 4: Atovaquone-proguanil
Started | 49 | 47 | 48 | 48
Completed | 29 | 27 | 32 | 32
Not Completed | 20 | 20 | 16 | 16
Not completed — Lack of Efficacy | 19 | 19 | 15 | 15
Not completed — OTHER: THE PARENT OF THE PARTICIPANT WHO IS A MINOR, WITHDREW THE PARTICIPANT FROM THE TRIAL | 1 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: M5717 (60 mg) + Pyronaridine | Cohort 2: M5717 (200 mg) + Pyronaridine | Cohort 3: M5717 (660 mg)+ Pyronaridine | Cohort 4: Atovaquone-proguanil | Total
Number analyzed (Participants) | 49 | 47 | 48 | 48 | 192
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23 (8.6) | 24 (8.9) | 25 (9.2) | 25 (11.2) | 25 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 20 | 19 | 75
  Male | 29 | 31 | 28 | 29 | 117
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity-Hispanic or Latino | 1 | 2 | 3 | 0 | 6
  Ethnicity-Not Hispanic or Latino | 48 | 45 | 44 | 48 | 185
  Ethnicity-Not Reported | 0 | 0 | 1 | 0 | 1
  Race-Black or African American | 49 | 47 | 48 | 48 | 192

OUTCOME MEASURES:

1. Primary Outcome: Time to Parasitemia Since Negative Blood Smear After Treatment
Description: The time (in days) to first recorded parasitemia (parasite count >0) since the first negative blood smear (parasite count of 0) after treatment (followed at least by 1 subsequent visit with a negative blood film), i.e. the time without a positive blood smear. Median time and 95% CI was estimated using the Kaplan Meier method for each cohort.
Time Frame: From treatment Day 1 up to End of observation period Day 64 (Week 10)
Population: The Full Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 1: M5717 (60 mg) + Pyronaridine | Cohort 2: M5717 (200 mg) + Pyronaridine | Cohort 3: M5717 (660 mg)+ Pyronaridine | Cohort 4: Atovaquone-proguanil
Number analyzed (Participants) | 49 | 47 | 48 | 48
days | 62.0 [49.0 to 100.0] | 60.0 [47.0 to 100.0] | NA [61.0 to 100.0] — Median not estimable due to an insufficient number of participants with events (parasitemia). | NA [59.0 to 100.0] — Median not estimable due to an insufficient number of participants with events (parasitemia).

2. Secondary Outcome: Percentage of Participants With Parasitemia (Positive Blood Smear)
Description: Percentage of participants with a positive blood smear (parasitemia) was reported. Parasitemia is the presence of parasites in blood (parasite count >0).
Time Frame: From treatment Day 1 up to End of observation period Day 64 (Week 10)
Population: The Full Analysis Set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: M5717 (60 mg) + Pyronaridine | Cohort 2: M5717 (200 mg) + Pyronaridine | Cohort 3: M5717 (660 mg)+ Pyronaridine | Cohort 4: Atovaquone-proguanil
Number analyzed (Participants) | 49 | 47 | 48 | 48
percentage of participants | 53.1 | 51.1 | 35.4 | 37.5

3. Secondary Outcome: Percentage of Participants With Polymerase Chain Reaction (PCR)-Adjusted Parasitemia (Due to New Infections)
Description: Percentage of participants with polymerase chain reaction (PCR)-adjusted Parasitemia (Thick Smear/Microscopy, after Adjustment for Parasitemia due to new Infections as determined by Genotyping using PCR Techniques) was reported.
Time Frame: From treatment Day 1 up to End of observation period Day 64 (Week 10)
Population: The Full Analysis Set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: M5717 (60 mg) + Pyronaridine | Cohort 2: M5717 (200 mg) + Pyronaridine | Cohort 3: M5717 (660 mg)+ Pyronaridine | Cohort 4: Atovaquone-proguanil
Number analyzed (Participants) | 49 | 47 | 48 | 48
percentage of participants | 40.8 | 36.2 | 29.2 | 31.3

4. Secondary Outcome: Percentage of Participants With PCR-adjusted Parasitemia (Due to Recrudescence)
Description: Percentage of participants with polymerase chain reaction (PCR)-adjusted Parasitemia (Thick Smear/Microscopy, after Adjustment for Parasitemia due to Recrudescence as determined by Genotyping using PCR Techniques) was reported.
Time Frame: From treatment Day 1 up to End of observation period Day 64 (Week 10)
Population: The Full Analysis Set included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: M5717 (60 mg) + Pyronaridine | Cohort 2: M5717 (200 mg) + Pyronaridine | Cohort 3: M5717 (660 mg)+ Pyronaridine | Cohort 4: Atovaquone-proguanil
Number analyzed (Participants) | 49 | 47 | 48 | 48
percentage of participants | 4.1 | 12.8 | 4.2 | 4.2

5. Secondary Outcome: Parasite Clearance Time
Description: Parasite clearance time defined as time from dosing to the first negative (no parasites) blood film (microscopy). Median parasite clearance time was estimated by Kaplan-Meier method
Time Frame: Time from dosing to the first negative (no parasites) blood film (microscopy) , assessed up to 12 weeks
Population: The Full Analysis Set included all randomized participants. Here overall number of participants analyzed signifies participants who had a baseline parasite density of >0.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Cohort 1: M5717 (60 mg) + Pyronaridine | Cohort 2: M5717 (200 mg) + Pyronaridine | Cohort 3: M5717 (660 mg)+ Pyronaridine | Cohort 4: Atovaquone-proguanil
Number analyzed (Participants) | 49 | 47 | 46 | 47
hours | 24.1 [6.2 to 39.0] | 24.2 [12.2 to 39.8] | 24.0 [12.1 to 48.2] | 25.0 [24.1 to 48.0]

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE), Serious TEAEs and Treatment Related TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered with study drug which does not necessarily had a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE was defined as AEs starting or worsening after the first intake of the study drug. TEAEs included both serious TEAEs and non-serious TEAEs. Treatment-related TEAEs: reasonably related to study intervention.
Time Frame: Up to End of Study (approximately 12 Weeks)
Population: Safety Analysis Set includes all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: M5717 (60 mg) + Pyronaridine | Cohort 2: M5717 (200 mg) + Pyronaridine | Cohort 3: M5717 (660 mg)+ Pyronaridine | Cohort 4: Atovaquone-proguanil
Number analyzed (Participants) | 49 | 47 | 48 | 48
Participants
  Participants with TEAEs | 31 | 27 | 31 | 28
  Participants with Serious TEAEs | 0 | 1 | 0 | 0
  Participants with Treatment-related TEAEs | 6 | 11 | 5 | 8

7. Secondary Outcome: Area Under the Blood Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M5717 and Pyronaridine
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUC extra represents an extrapolated value obtained by Clast/ λz, where Clast is the calculated blood concentration at the last sampling time point at which the measured blood concentration is at or above the Lower Limit of quantification (LLQ) and λz is the apparent terminal rate constant determined by log-linear regression analysis of the measured blood concentrations of the terminal log-linear phase.
Time Frame: Predose, 1, 2, 4, 6, 8, and 12 hours on Day 1 and 24 hours on Day 2
Population: Pharmacokinetic (PK) analysis set included all participants, who received 1 dose of M5717, had no clinically important protocol deviations/important events affecting PK, & provide at least 1 measurable post-dose concentration. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter(hour*ng/mL)
Groups:
- Cohort 1: M5717 60 mg: Participants received a single oral dose of M5717 60 milligrams (mg) once daily in a single-day treatment regimen on Day 1 under fasting condition.
- Cohort 2: M5717 200 mg: Participants received a single oral dose of M5717 200 milligrams (mg) in a single-day treatment regimen administered under fasting conditions on Day 1 under fasting condition.
- Cohort 3: M5717 660 mg: Participants received a single oral dose of M5717 660 mg as part of a single-day treatment regimen on Day 1 under fasting condition.
- Cohort 1, 2 and 3: Pyronaridine 540 mg: Participants received a single pyronaridine tetraphosphate (pyronaridine) 540 mg for those weighing between ≥ 45 kg and < 65 kg-in a single-day treatment regimen administered under fasting conditions on Day 1 under fasting condition in Cohorts 1, 2 and 3.
- Cohort 1, 2 and 3: Pyronaridine 720 mg: Participants received 720 mg for those weighing ≥ 65 kilograms (kg) as part of a single-day treatment regimen on Day 1 under fasting condition in Cohorts 1, 2 and 3.
Arm/Group | Cohort 1: M5717 60 mg | Cohort 2: M5717 200 mg | Cohort 3: M5717 660 mg | Cohort 1, 2 and 3: Pyronaridine 540 mg | Cohort 1, 2 and 3: Pyronaridine 720 mg
Number analyzed (Participants) | 45 | 44 | 43 | 99 | 33
hour*nanogram per milliliter(hour*ng/mL) | 613.64 (1.1) | 2292.02 (0.5) | 9988.92 (0.4) | 5985.14 (0.5) | 6418.17 (0.3)

8. Secondary Outcome: Area Under the Blood Concentration-Time Curve From Time Zero to 24 Hours Post-dose (AUC 0-24) of M5717 and Pyronaridine
Description: AUC from time zero to 24 hours post dose, calculated using the mixed log linear trapezoidal rule (linear up, log down) using the nominal dosing interval.
Time Frame: Predose, 1, 2, 4, 6, 8, and 12 hours on Day 1 and 24 hours on Day 2
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- M5717 60 mg: Participants received a single oral dose of M5717 60 milligrams (mg) once daily in a single-day treatment regimen on Day 1 under fasting condition.
Arm/Group | M5717 60 mg | Cohort 2: M5717 200 mg | Cohort 3: M5717 660 mg | Cohort 1, 2 and 3: Pyronaridine 540 mg | Cohort 1, 2 and 3: Pyronaridine 720 mg
Number analyzed (Participants) | 45 | 44 | 43 | 99 | 33
h*ng/mL | 205.87 (0.4) | 743.74 (0.5) | 3303.65 (0.4) | 1594.05 (0.6) | 1742.89 (0.4)

9. Secondary Outcome: Area Under the Blood Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC 0-tlast) of M5717 and Pyronaridine
Description: Area under the blood concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Predose, 1, 2, 4, 6, 8, and 12 hours on Day 1 and 24 hours on Day 2
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Cohort 3: M5717 (660 mg): Participants received a single oral dose of M5717 660 mg as part of a single-day treatment regimen on Day 1 under fasting condition.
Arm/Group | Cohort 1: M5717 60 mg | Cohort 2: M5717 200 mg | Cohort 3: M5717 (660 mg) | Cohort 1, 2 and 3: Pyronaridine 540 mg | Cohort 1, 2 and 3: Pyronaridine 720 mg
Number analyzed (Participants) | 45 | 44 | 43 | 99 | 33
h*ng/mL | 455.40 (0.5) | 2040.41 (0.5) | 9635.73 (0.4) | 5393.62 (0.6) | 5793.71 (0.4)

10. Secondary Outcome: Apparent Total Body Clearance From Blood (CL/f) of M5717 and Pyronaridine
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent body clearance of the drug from blood, CL= Dose/AUC0-inf.
Time Frame: Predose, 1, 2, 4, 6, 8, and 12 hours on Day 1 and 24 hours on Day 2
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per Hours (L/h)
Arm/Group | Cohort 1: M5717 60 mg | Cohort 2: M5717 200 mg | Cohort 3: M5717 660 mg | Cohort 1, 2 and 3: Pyronaridine 540 mg | Cohort 1, 2 and 3: Pyronaridine 720 mg
Number analyzed (Participants) | 45 | 44 | 43 | 99 | 33
Liter per Hours (L/h) | 97.77 (1.1) | 87.25 (0.5) | 66.07 (0.4) | 90.22 (0.5) | 112.18 (0.3)

11. Secondary Outcome: Maximum Observed Blood Concentration (Cmax) of M5717 and Pyronaridine
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Predose, 1, 2, 4, 6, 8, and 12 hours on Day 1 and 24 hours on Day 2
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: M5717 60 mg | Cohort 2: M5717 200 mg | Cohort 3: M5717 660 mg | Cohort 1, 2 and 3: Pyronaridine 540 mg | Cohort 1, 2 and 3: Pyronaridine 720 mg
Number analyzed (Participants) | 45 | 44 | 43 | 99 | 33
nanogram per milliliter (ng/mL) | 15.19 (0.6) | 59.69 (0.6) | 254.50 (0.5) | 157.81 (0.6) | 166.46 (0.4)

12. Secondary Outcome: Apparent Terminal Half-life (t1/2) of M5717 and Pyronaridine
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by lambda z.
Time Frame: Predose, 1, 2, 4, 6, 8, and 12 hours on Day 1 and 24 hours on Day 2
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Cohort 1: M5717 60 mg | Cohort 2: M5717 200 mg | Cohort 3: M5717 660 mg | Cohort 1, 2 and 3: Pyronaridine 540 mg | Cohort 1, 2 and 3: Pyronaridine 720 mg
Number analyzed (Participants) | 45 | 44 | 43 | 99 | 33
hour | 46.013 (1.3) | 64.663 (0.4) | 90.234 (0.5) | 264.15 (0.4) | 246.94 (0.6)

13. Secondary Outcome: Time to Reach the Maximum Blood Concentration (Tmax) of M5717 and Pyronaridine
Description: Time to reach the maximum blood concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Predose, 1, 2, 4, 6, 8, and 12 hours on Day 1 and 24 hours on Day 2
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: M5717 60 mg | Cohort 2: M5717 200 mg | Cohort 3: M5717 660 mg | Cohort 1, 2 and 3: Pyronaridine 540 mg | Cohort 1, 2 and 3: Pyronaridine 720 mg
Number analyzed (Participants) | 45 | 44 | 43 | 99 | 33
hour | 4.067 [1.05 to 141.07] | 4.00 [1.00 to 12.10] | 4.00 [1.08 to 175.57] | 2.10 [1.00 to 7.42] | 2.08 [1.00 to 12.08]

14. Secondary Outcome: Apparent Volume of Distribution (Vz/F) During the Terminal Phase of M5717 and Pyronaridine
Description: The Vz/f was defined as the theoretical volume in which the total amount of required to uniformly distribute to produce the desired plasma concentration. Apparent volume of distribution after oral dose (Vz/F) was influenced by the fraction absorbed. The Vz/f was calculated by dividing the dose with area under the concentration time curve from time zero to infinity multiplied with terminal elimination rate constant Lambda(z). Vz/f=Dose/AUC(0-inf) multiply Lambda(z).
Time Frame: Predose, 1, 2, 4, 6, 8, and 12 hours on Day 1 and 24 hours on Day 2
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Cohort 1: M5717 60 mg | Cohort 2: M5717 200 mg | Cohort 3: M5717 660 mg | Cohort 1, 2 and 3: Pyronaridine 540 mg | Cohort 1, 2 and 3: Pyronaridine 720 mg
Number analyzed (Participants) | 45 | 44 | 43 | 99 | 33
liter | 6490.76 (0.5) | 8140.36 (0.4) | 8601.43 (0.5) | 34383.091 (0.5) | 39966.70 (0.7)

ADVERSE EVENTS:
Time Frame: End of Study (approximately 12 Weeks)
Arm/Group | Cohort 1: M5717 (60 mg) + Pyronaridine | Cohort 2: M5717 (200 mg) + Pyronaridine | Cohort 3: M5717 (660 mg)+ Pyronaridine | Cohort 4: Atovaquone-proguanil
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/47 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/47 | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 31/49 | 27/47 | 31/48 | 28/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: M5717 (60 mg) + Pyronaridine (N=49) | Cohort 2: M5717 (200 mg) + Pyronaridine (N=47) | Cohort 3: M5717 (660 mg)+ Pyronaridine (N=48) | Cohort 4: Atovaquone-proguanil (N=48)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: M5717 (60 mg) + Pyronaridine (N=49) | Cohort 2: M5717 (200 mg) + Pyronaridine (N=47) | Cohort 3: M5717 (660 mg)+ Pyronaridine (N=48) | Cohort 4: Atovaquone-proguanil (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 14 (14) | 12 (12) | 10 (10) | 7 (7)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasmodium ovale infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Schistosomiasis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (4) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 3 (3) | 2 (2) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 5 (5) | 6 (6) | 3 (3) | 7 (7)
Blood bilirubin increased (Investigations) | 7 (7) | 4 (4) | 4 (4) | 4 (4)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Monocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pH urine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Red blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypercreatininaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 7 (7) | 3 (3) | 6 (6) | 9 (9)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT05974267/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT05974267/SAP_001.pdf